CLINICAL TRIAL: NCT01087736
Title: Topiramate Treatment of Alcohol Use Disorders in Veterans With Post Traumatic Stress Disorder (PTSD): A Pilot Controlled Trial of Augmentation Therapy
Acronym: TAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H5220-34690-01; DAMD17-03-1-0532 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: PTSD; Alcohol Abuse; Alcoholism
Keywords: PTSD; Alcohol abuse; Alcoholism; Topiramate; Stress Disorder, Post Traumatic; Chronic Post-Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism | interventions — Topiramate; Qnexa; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topiramate (Experimental): Participants will be randomly assigned to either the topiramate arm or placebo arm. Neither the participant nor the researchers will know which arm the participant is in. Participants in the topiramate arm will be ingesting daily doses of topiramate that will gradually increase to a maximum, and then taper off.
  Interventions: Drug: Topiramate
- Placebo (Placebo Comparator): The Drug Product Services Laboratory at UCSF will purchase and supply our lab with USP or NF grade topiramate study capsules and matching placebo capsules. Randomization will be done by a consulting biostatistician, who will be the only one to know which participants are assigned to placebo. Dosing will follow the same procedures as with topiramate in that arm of the study. If adverse events occur, there will be a procedure in place for unblinding only that participant.
  Interventions: Other: Placebo administration

INTERVENTIONS:
Drug: Topiramate — After random assignment, topiramate will be titrated up over 5 weeks. Dosing begins at 25 mg per day, and increase in the second week to 25 mg twice per day; in the third week to 50 mg twice/day; in the fourth week to 75 mg twice/day; in the 5th week to 100 mg twice/day; and in weeks 6-11 increased to and maintained at 100 mg in the morning and 200 mg at night. Patients will receive the highest dose tolerated, not to exceed 300 mg per day. Adjustments are permitted throughout titration. Once maximum tolerated dosage is reached, subjects will be asked to maintain dosage for remainder of the treatment phase. Upon completing the 6 week maintenance period subjects will taper off over a 7-day period (Week 12). If subjects experience significant side effects, the dosage may be adjusted.
  Other Names: Topamax; Qnexa
  Arms: Topiramate
Other: Placebo administration — Placebo pills will be prepared by the UCSF pharmacy which will be indistinguishable from the topiramate pills used in that arm. Both topiramate and placebo will then be delivered to the VA pharmacy. A consulting biostatistician will randomly assign participants to either the topiramate or placebo group. The dosing of placebo pills will follow the same regimen as outlined for the topiramate arm. In the event of a safety issue, there will be a procedure for unblinding only that participant.
  Other Names: Placebo; Sugar pill
  Arms: Placebo

SUMMARY:
The proposed project aims to:

1. Obtain a preliminary assessment of the efficacy of topiramate treatment in reducing alcohol use in veterans with Post Traumatic Stress Disorder (PTSD) and alcohol dependence;
2. Obtain preliminary assessments of safety/tolerability of topiramate in these patients;
3. Assess the feasibility of recruitment and retention for topiramate treatment in this comorbid population; and 4) to inform the design of a planned subsequent larger controlled trial of topiramate.

PRIMARY HYPOTHESIS: Topiramate treatment combined with Medical Management alcohol counseling will be associated with a significant decrease in percent drinking days from baseline to end of treatment.

SECONDARY HYPOTHESIS: There will be significantly less percent drinking days in the topiramate treatment group compared to the placebo group.

DETAILED DESCRIPTION:
The goal of the proposed project is to improve the treatment of veterans with co-occurring Post Traumatic Stress Disorder (PTSD) and alcohol dependence. Exposure to the stresses of combat is known to be associated with risk for both PTSD and alcohol and other substance use. PTSD and alcohol use disorders occur frequently among returning OEF/OIF veterans. Alcohol and substance use are risk factors for the development of PTSD, moderators of PTSD symptom severity, and potential consequences of PTSD. Alcohol is by far the most common substance of abuse in patients with PTSD, and its use may represent an attempt by PTSD patients to "self-medicate" symptoms such as hyperarousal. However, to date there has been little research to develop pharmacotherapies that would, ideally, reduce both alcohol use and PTSD symptoms.

Topiramate is one of the few medications for alcohol dependence that has also been tested as a potential medication to treat PTSD. Topiramate's efficacy in alcohol dependence has been shown in two recent large controlled trials. Several open trials have suggested that topiramate may be effective in reducing PTSD symptoms while the results of two small controlled trials have been mixed.

A clinical trial of topiramate is therefore indicated in order to achieve the following specific aims:

The primary aim is to obtain a preliminary assessment of the efficacy of topiramate in increasing the percent of days abstinent from alcohol use from baseline to the end of treatment in veterans with PTSD and alcohol abuse/dependence who are drinking heavily.

The secondary aim is to obtain a preliminary assessment of the efficacy of topiramate in increasing the percent of days abstinent from alcohol as compared to placebo.

Additional aims include the following:

* To obtain a preliminary assessment of the efficacy of topiramate in reducing other measures of alcohol use such as percent heavy drinking days, number of drinks per week, number of drinks per drinking day, and alcohol craving.
* To obtain a preliminary assessment of the efficacy of topiramate in reducing PTSD symptom severity in veterans with chronic PTSD and alcohol abuse/dependence.
* Informing the design of a planned subsequent larger controlled trial of topiramate in veterans with chronic PTSD and alcohol abuse/dependence
* To obtain an estimate of topiramate vs. placebo effect size for future studies. B. To obtain a preliminary assessment of the effects of topiramate treatment on measures of risk-taking behavior in veterans with chronic PTSD and alcohol abuse/dependence.

To achieve these aims, we will conduct a prospective, parallel groups, randomized, double-blind, placebo-controlled flexible-dose pilot clinical trial of topiramate in veterans with PTSD and alcohol abuse/dependence who are already receiving standard treatment for PTSD but still drink heavily. The primary treatment outcome will be percent days abstinent from alcohol; secondary outcomes will include other alcohol use measures, PTSD symptom severity, adverse effects, recruitment and retention rates.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatient veterans.
* Current DSM-IV diagnosis of PTSD.
* Current (past month) DSM-IV diagnosis of an Alcohol Use Disorder.
* Must meet criteria for "heavy" or "at-risk" drinking by NIAAA thresholds.
* Receiving treatment for PTSD.
* Must express desire to reduce alcohol consumption.
* Female subjects must have negative urine pregnancy test and must be either postmenopausal for at least one year, or practicing an effective method of birth control.
* Must have a BAC of less than 0.02% when signing the informed consent.

Exclusion Criteria:

* Psychotic disorders, bipolar disorder, dementia, or other psychiatric disorders judged to be unstable.
* Subjects known to have clinically significant unstable medical conditions, including but not limited to: clinically significant renal disease and/or impaired renal function as defined by clinically significant elevation of BUN or creatinine or an estimated creatinine clearance of < 60 mL/min; AST (SGOT) and/or ALT (SGPT) >3 times the upper limit of the normal range and/or an increased serum bilirubin >2 times the upper limit of normal; seizure disorders.
* Subjects with glaucoma.
* Subjects with a history of kidney stones.
* Subjects with a history of renal disease.
* Concurrent participation in another treatment study.
* Female patients who are pregnant or lactating.
* Current topiramate use or use within the past 4 weeks.
* Current medications for alcohol dependence or use within the past 4 weeks.
* Needing acute medical detoxification from alcohol based on a score of 12 or more on the Clinical Institute Withdrawal Assessment of Alcohol Scale (CIWA-AD);
* Subjects who are legally mandated to participate in an alcohol treatment program.
* Subjects who have had a suicide attempt or suicidal ideation in the 6 months prior to enrollment.
* Subjects who have previously been treated with topiramate for any reason and discontinued treatment due to an adverse event or due to a hypersensitivity reaction to topiramate,
* Subjects with seizure disorders that require anticonvulsant medications
* Subjects currently being treated with another anticonvulsant.
* Subjects who in the opinion of the investigator should not be enrolled in the study because of the precautions,warnings or contraindications outlined in the topiramate package insert.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-04; Primary Completion 2012-09 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven L. Batki, MD, Principal Investigator — University of California, San Francisco; Department of Veteran's Affairs
Locations (1):
- San Francisco VA Medical Center, San Francisco, California, United States

REFERENCES:
- [Background] Alderman CP, McCarthy LC, Condon JT, Marwood AC, Fuller JR. Topiramate in combat-related posttraumatic stress disorder. Ann Pharmacother. 2009 Apr;43(4):635-41. doi: 10.1345/aph.1L578. Epub 2009 Mar 31. PMID 19336652
- [Background] Anton RF, O'Malley SS, Ciraulo DA, Cisler RA, Couper D, Donovan DM, Gastfriend DR, Hosking JD, Johnson BA, LoCastro JS, Longabaugh R, Mason BJ, Mattson ME, Miller WR, Pettinati HM, Randall CL, Swift R, Weiss RD, Williams LD, Zweben A; COMBINE Study Research Group. Combined pharmacotherapies and behavioral interventions for alcohol dependence: the COMBINE study: a randomized controlled trial. JAMA. 2006 May 3;295(17):2003-17. doi: 10.1001/jama.295.17.2003. PMID 16670409
- [Background] Anton RF, Moak DH, Latham P. The Obsessive Compulsive Drinking Scale: a self-rated instrument for the quantification of thoughts about alcohol and drinking behavior. Alcohol Clin Exp Res. 1995 Feb;19(1):92-9. doi: 10.1111/j.1530-0277.1995.tb01475.x. PMID 7771669
- [Background] Baker F, Johnson MW, Bickel WK. Delay discounting in current and never-before cigarette smokers: similarities and differences across commodity, sign, and magnitude. J Abnorm Psychol. 2003 Aug;112(3):382-92. doi: 10.1037/0021-843x.112.3.382. PMID 12943017
- [Background] Batki SL, Dimmock JA, Wade M, Gately PW, Cornell M, Maisto SA, Carey KB, Ploutz-Snyder R. Monitored naltrexone without counseling for alcohol abuse/dependence in schizophrenia-spectrum disorders. Am J Addict. 2007 Jul-Aug;16(4):253-9. doi: 10.1080/10550490701389732. PMID 17661192
- [Background] Beckham JC, Crawford AL, Feldman ME. Trail making test performance in Vietnam combat veterans with and without posttraumatic stress disorder. J Trauma Stress. 1998 Oct;11(4):811-9. doi: 10.1023/A:1024409903617. PMID 9870231
- [Background] Berlant J, van Kammen DP. Open-label topiramate as primary or adjunctive therapy in chronic civilian posttraumatic stress disorder: a preliminary report. J Clin Psychiatry. 2002 Jan;63(1):15-20. doi: 10.4088/jcp.v63n0104. PMID 11838620
- [Background] Berlant JL. Prospective open-label study of add-on and monotherapy topiramate in civilians with chronic nonhallucinatory posttraumatic stress disorder. BMC Psychiatry. 2004 Aug 18;4:24. doi: 10.1186/1471-244X-4-24. PMID 15315714

RESULTS

PARTICIPANT FLOW:
Groups:
- Topiramate: Topiramate: topiramate titrated up over 5 weeks, beginning at 25 mg per day, and increased in the second week to 25 mg twice per day; in the third week to 50 mg twice/day; in the fourth week to 75 mg twice/day; in the 5th week to 100 mg twice/day; and in weeks 6-11 increased to and maintained at 100 mg in the morning and 200 mg at night. Upon completing the 6 week maintenance period dosage was tapered off over a 7-day period (Week 12).
- Placebo: Placebo: Placebo pills prepared by the UCSF pharmacy were indistinguishable from the topiramate pills used in that arm. The dosing of placebo pills followed the same regimen as outlined for the topiramate arm. In the event of a safety issue, there would be a procedure for unblinding only that participant.
Period: Overall Study
Arm/Group | Topiramate | Placebo
Started | 14 | 16
Completed | 13 | 14
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topiramate | Placebo | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (13.9) | 50.4 (12.8) | 50 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 13 | 15 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 5 | 7
  White | 8 | 8 | 16
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 16 | 30
History of combat exposure [Number; unit: participants]
  Combat exposure | 10 | 12 | 22
  No combat exposure | 4 | 4 | 8
Comorbid substance use disorder [Number; unit: participants]
  Comorbid substance use disorder present | 5 | 5 | 10
  Comorbid substance use disorder absent | 9 | 11 | 20
Prior treatment for substance use disorder [Number; unit: participants]
  Residential treatment | 4 | 2 | 6
  Outpatient treatment | 7 | 8 | 15
  No prior substance use disorder treatment | 3 | 6 | 9
BDI [Mean (Standard Deviation); unit: units on a scale] — Depression was assessed using the Beck Depression Inventory, scores range from 0-63, with scores over 40 indicating severe depression and scores under 10 indicating normal mood symptoms.
  units on a scale | 23.4 (11.6) | 26.3 (12.3) | 24.9 (11.9)
BAI [Mean (Standard Deviation); unit: units on a scale] — The Beck Anxiety Inventory (BAI) consists of twenty-one questions about how the subject has been feeling in the last week, expressed as common symptoms of anxiety (such as numbness and tingling, sweating not due to heat, and fear of the worst happening).Each question has the same set of four possible answer choices, ranging from 0 to 3 points: NOT AT ALL (0), MILDLY (1), MODERATELY (2), SEVERELY (3). Total BAI scores range from 0 - 63, with higher scores indicating greater severity.
  0-7: minimal level of anxiety 8-15: mild anxiety 16-25: moderate anxiety 26-63: severe anxiety
  units on a scale | 20.4 (12.7) | 27.4 (13.3) | 24.0 (13.3)
Alcohol Use Disorders Identification Test [Mean (Standard Deviation); unit: units on a scale] — The Alcohol Use Disorders Identification Test (AUDIT) score is the sum of 10 questions about alcohol consumption, each with scores ranging from 0 to 4, and total AUDIT score ranges from 0-40. Higher scores indicate greater likelihood of hazardous and harmful drinking, and may also reflect greater severity of alcohol problems and dependence, as well as a greater need for more intensive treatment.
  units on a scale | 27.1 (7.9) | 23.0 (7.5) | 24.9 (7.8)
Percent drinking days per week [Mean (Standard Deviation); unit: percent days in a week] — The Alcohol Timeline Followback (TLFB) is a drinking assessment interview that obtains estimates of daily drinking and has been evaluated with clinical and nonclinical populations. Using a calendar, people provided retrospective estimates of their daily drinking over the 90 day period prior to study screening.
  DD: day on which alcohol was consumed
  percent days in a week | 73.3 (30.3) | 80.4 (21.5) | 77.1 (25.8)
Percent heavy drinking days per week [Mean (Standard Deviation); unit: percent days in a week] — The Alcohol Timeline Followback (TLFB) is a drinking assessment interview that obtains estimates of daily drinking and has been evaluated with clinical and nonclinical populations. Using a calendar, people provided retrospective estimates of their daily drinking over the 90 day period prior to study screening.
  HDD: day on which >4 (men) or >3 (women) standard alcoholic drinks were consumed Standard alcoholic drink defined as containing 13.6 g of pure alcohol.
  percent days in a week | 58.5 (33.7) | 72.6 (28.5) | 66.0 (31.3)
Average drinks per week [Mean (Standard Deviation); unit: Drinks] — The Alcohol Timeline Followback (TLFB) is a drinking assessment interview that obtains estimates of daily drinking and has been evaluated with clinical and nonclinical populations. Using a calendar, people provided retrospective estimates of their daily drinking over the 90 day period prior to study screening.
  Standard alcoholic drink defined as containing 13.6 g of pure alcohol.
  Drinks | 52.4 (34.2) | 58.2 (25.4) | 55.5 (29.4)
Average drinks per drinking day [Mean (Standard Deviation); unit: Drinks] — The Alcohol Timeline Followback (TLFB) is a drinking assessment interview that obtains estimates of daily drinking and has been evaluated with clinical and nonclinical populations. Using a calendar, people provided retrospective estimates of their daily drinking over the 90 day period prior to study screening.
  DD: day on which alcohol was consumed Standard alcoholic drink defined as containing 13.6 g of pure alcohol.
  Drinks | 11.1 (6.1) | 10.9 (4.7) | 11.0 (5.3)
Baseline PTSD Symptomatology [Mean (Standard Deviation); unit: units on a scale] — The Clinician-Administered PTSD Checklist (CAPS) was used at baseline to assess PTSD symptoms at baseline. The PTSD Checklist is a measure of the 17 DSM-IV symptoms of PTSD. Respondents rate on a scale from 1 (not at all) to 5 (extremely) how much they were bothered by each symptom in the past month. A total symptom severity score (range = 17 - 85) can be obtained by summing the scores from the 17 items, with higher scores indicating greater severity of PTSD symptoms. Mean scores may be calculated for subscales of intrusion (range 5-25), avoidance (range 7-35), and arousal (range 5-25).
  units on a scale
    PTSD total score | 72.8 (14.3) | 83.1 (17.3) | 78.3 (16.6)
    Intrusion subscale | 18.2 (4.3) | 21.9 (6.9) | 20.2 (6.0)
    Avoidance subscale | 31.1 (6.1) | 34.8 (8.9) | 33.1 (7.8)
    Arousal subscale | 23.5 (6.7) | 26.4 (4.1) | 25.0 (5.6)

OUTCOME MEASURES:

1. Primary Outcome: Percent Drinking Days (%DD)
Description: Alcohol consumption was assessed at baseline and weekly during the treatment phase (12 weeks) using the Time Line Follow Back (TLFB) interview which yields number of days of alcohol use (DD).
  DD: day on which alcohol was consumed Standard alcoholic drink defined as containing 13.6 g of pure alcohol.
Time Frame: Weekly, weeks 1-12, average
Measure: Mean (Standard Deviation); unit: percent days in a week
Arm/Group | Topiramate | Placebo
Number analyzed (Participants) | 14 | 16
percent days in a week | 19.5 (34.2) | 39.7 (36.5)
Statistical Analysis 1: Comparison: Topiramate; Our primary protocol-defined analysis was to examine the within-group efficacy of topiramate to reduce percent drinking days (%DD); Test type: Superiority or Other; p = 0.019, negative binomial regression — We tested our Primary hypothesis with a random-intercept repeated subject negative binomial model, modeling week (baseline - week 12) as a continuous variable. All analyses were intent-to-treat and used all observations from all weeks; Incidence Rate Ratio (IRR) = 0.89, 95% CI 2-sided [0.89 to 0.98]
Statistical Analysis 2: Comparison: Placebo; There were no pre hoc hypothesis regarding change within placebo group. We were only tested change within the topiramate condition; Test type: Superiority or Other; p = 0.00, Other
Statistical Analysis 3: Comparison: Topiramate vs Placebo; A secondary analysis was powered to detect a "Signal" or statistical trend (p<0.10) for a difference between the topiramate and placebo condition. We compared percent drinking days per week between groups averaged over the active phase of the trial (weeks 1-12). The negative binomial model included fixed effect for week, treatment group, and the interaction between treatment group and week. We covaried for baseline %DD averages to control for prestudy and study enrollment effects; Test type: Superiority or Other; p = 0.036, Negative binomial model; Incidence Rate Ratio (IRR) = 0.38, 95% CI 2-sided [0.15 to 0.94]

2. Other Pre Specified Outcome: PTSD Symptom Severity
Description: The average PTSD symptom severity score during treatment (weeks 4, 8, 12). The PTSD Checklist (PCL) is a self-report measure of the 17 DSM-IV symptoms of PTSD. Respondents rate on a scale from 1 (not at all) to 5 (extremely) how much they were bothered by each symptom in the past month. A total symptom severity score (range = 17 - 85) can be obtained by summing the scores from the 17 items, with higher scores indicating greater severity of PTSD symptoms. Mean scores may be calculated for subscales of intrusion (range 5-25), avoidance (range 7-35), and arousal (range 5-25).
Time Frame: Weeks 4, 8, 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Topiramate | Placebo
Number analyzed (Participants) | 14 | 16
units on a scale
  PCL Total Score (Weeks 1-12 Average) | 42.3 (16.4) | 49.0 (16.5)
  PCL-B Intrusion (Weeks 1-12 Average) | 12.3 (5.5) | 14.3 (5.5)
  PCL-C Avoidance (Weeks 1-12 Average) | 17.6 (7.4) | 19.9 (6.9)
  PCL-D Arousal (Weeks 1-12 Average) | 12.4 (4.9) | 14.9 (5.0)
Statistical Analysis 1: Comparison: Topiramate; We planned to explore the efficacy of topiramate in reducing PTSD symptom severity. We used random-intercept linear mixed models to explore the efficacy for topiramate related reduction in PTSD symptomatology. We looked for an effect of week within TOP. Baseline scores for PTSD symptoms were used as covariates in group comparisons. All analyses were intent-to-treat and used all observations from all weeks; Test type: Superiority or Other; p < 0.026, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo; There was not a pre hoc hypothesis regarding change within placebo group. We only examined within group change in the topiramate condition; Test type: Superiority or Other; p = 0.00, Other

ADVERSE EVENTS:
Time Frame: 12 Weeks
Arm/Group | Topiramate | Placebo
Serious Adverse Events (participants affected / at risk) | 0/14 | 4/16
Other Adverse Events (participants affected / at risk) | 12/14 | 13/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topiramate (N=14) | Placebo (N=16)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) — Subject was hospitalized due to alcohol relapse and self-reported suicidal ideation
Chest pain (Cardiac disorders) | 0 (0) | 2 (4) — Myocardial infarction (MI) was ruled out and patient was discharged the next day
Death (General disorders) | 0 (0) | 1 (1) — Research participant in 9th week of treatment died of apparent cardiac arrest
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topiramate (N=14) | Placebo (N=16)
numbness/tingling (Nervous system disorders) | 3 (3) | 2 (2)
Altered taste (Nervous system disorders) | 3 (3) | 5 (5)
Difficulty with concentration/attention (Nervous system disorders) | 2 (2) | 1 (1)
Difficulty with memory (Nervous system disorders) | 1 (1) | 1 (1)
Slow thinking (Nervous system disorders) | 2 (2) | 2 (2)
Confusion (Nervous system disorders) | 2 (2) | 3 (3)
Language problems (Nervous system disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 3 (3) | 2 (2)
Loss of appetite (General disorders) | 4 (4) | 6 (6)
Dizziness (General disorders) | 1 (1) | 4 (4)
Itching (General disorders) | 3 (3) | 1 (1)
Sleepiness (General disorders) | 5 (5) | 2 (2)
Nervousness (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 3 (3)
Abnormal vision (Eye disorders) | 3 (3) | 3 (3)
Eye pain (Eye disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes